CLINICAL TRIAL: NCT00004664
Title: Randomized Placebo-Controlled Study of Aerobic Exercise and Resistance Training Plus Megestrol Acetate for HIV-Wasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11931; NU-516
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Wasting Syndrome; HIV Infections
Keywords: disease-related problem/condition; human immunodeficiency virus infection; immunologic disorders and infectious disorders; nutrition; rare disease; viral infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Wasting Syndrome; HIV Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Megestrol; Exercise

INTERVENTIONS:
Drug: megestrol
Behavioral: Exercise

SUMMARY:
OBJECTIVES: I. Evaluate the effect of aerobic exercise and progressive resistance plus megestrol acetate on lean body mass of patients with human immunodeficiency virus-related weight loss (HIV-wasting).

II. Evaluate whether exercise acutely alters immune function. III. Evaluate whether long-term exercise improves immunocompetence. IV. Evaluate the accuracy of multifrequency bioelectrical impedance spectral analysis in measuring body composition.

V. Assess the impact of these therapies on quality of life. VI. Evaluate the effect of these therapies on the balance of energy intake and energy expenditure.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are randomly assigned to 1 of 3 therapy groups: megestrol acetate alone, exercise plus megestrol acetate, or exercise plus placebo. Therapy continues for 12 weeks.

A single dose of oral megestrol acetate or placebo is administered each morning.

The exercise program consists of aerobic exercise and resistance training performed 3 times a week under supervision. Hard aerobic exercise is performed for 45 minutes plus a warm-up and cool-down period; the patient chooses to work on 3 of 5 pieces of exercise equipment. Exercise intensity is adjusted to a heart rate corresponding to 65% of maximal oxygen consumption.

Resistance training is done on a universal gym; exercises are designed to work all 6 major muscle groups. Each exercise is performed at 70% of maximal single repetition resistance. Resistance is increased 5% when the patient can perform 15 repetitions without failure.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Human immunodeficiency virus seropositive with acquired immune deficiency syndrome

Documented weight loss 5% to 15% below ideal weight

--Prior/Concurrent Therapy--

No concurrent appetite stimulants

At least 6 weeks since initiation of new antiretroviral therapy

--Patient Characteristics--

Performance status: Karnofsky 70%-100%

Hepatic: No ascites

Renal: No nephrosis

Other:

* No acute or untreated infection within 4 weeks prior to entry
* No hospitalization within 2 weeks prior to entry
* No gonadal insufficiency
* No edema
* No pleural effusion
* No uncontrolled diarrhea
* No physical or functional obstruction to food intake
* No physical handicap that would prevent resistance or aerobic exercise
* No cardiac abnormality that would render aerobic exercise a health risk
* No concurrent regular exercise of 3 or more hours a week
* No mental incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hayden Von Roenn, Study Chair — Northwestern University